CLINICAL TRIAL: NCT06369298
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of JK07 in Adults With Chronic Heart Failure (RENEU-HF)
Brief Title: Study of JK07 in Patients With Chronic Heart Failure
Acronym: RENEU-HF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Salubris Biotherapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JK07.2.01
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Heart Failure with Reduced Ejection Fraction; Heart Failure with Preserved Ejection Fraction; Heart Failure NYHA Class III; Heart Failure NYHA Class II; Heart Failure with Atrial Fibrillation/Flutter; HFrEF; HFpEF; Neuregulin 1; NRG-1; HER3; HER4; ErbB3; ErbB4; Systolic Heart Failure; Diastolic Heart Failure; Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Heart Failure; Fibromatosis, Gingival, 2; Heart Failure, Systolic; Heart Failure, Diastolic; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- JK07 low dose (Active Comparator): JK07 administered by intravenous (IV) infusion
  Interventions: Drug: JK07
- JK07 high dose (Active Comparator): JK07 administered by intravenous (IV) infusion
  Interventions: Drug: JK07
- Placebo (Placebo Comparator): Placebo administered by intravenous (IV) infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JK07 — JK07 is a fully human anti-human epidermal growth factor receptor 3 (also known as ErbB3 or HER3) antibody fused with the epidermal growth factor (EGF)-domain of Neuregulin (NRG)-1b protein.
  Arms: JK07 high dose; JK07 low dose
Drug: Placebo — 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, multiple dose study to assess the safety, tolerability, and efficacy of JK07 in participants aged 18-85 with heart failure.

There will be 2 cohorts in this study:

Cohort 1: Heart failure (HF) participants with left ventricular ejection fraction (LVEF) of ≤ 40%.

Cohort 2: Heart failure (HF) participants with left ventricular ejection fraction (LVEF) > 40% and ≤ 65%.

ELIGIBILITY:
Inclusion Criteria:

* Participants with New York Heart Association (NYHA) Class II-III.
* Cohort 1 - Left Ventricular Ejection Fraction (LVEF) ≤ 40%.
* Cohort 2 - Left Ventricular Ejection Fraction (LVEF) >40% and ≤ 65%, elevated N-terminal pro B-type natriuretic peptide (NT-proBNP) ≥ 600pg/mL and atrial fibrillation/flutter.
* Stable heart failure and on optimal medical therapy.
* Screening hemoglobin ≥ 9.0 g/dL.

Exclusion Criteria:

* Uncontrolled hypertension.
* Sustained systolic Blood Pressure (BP) < 90 mmHg and/or diastolic BP < 50 mmHg on 2 consecutive (duplicate seated) readings at screening.
* Heart failure due to hypertrophic cardiomyopathy, restrictive and/or infiltrative cardiomyopathy, arrhythmogenic right ventricular dysplasia, Fabry disease, or Noonan syndrome with LV hypertrophy or a positive serum immunofixation result.
* Diagnosis of stress-induced (Takotsubo) cardiomyopathy, myocarditis, or peripartum cardiomyopathy.
* Diagnosis of chemotherapy- or radiation-induced cardiomyopathy.
* Diagnosed with stroke or Transient Ischemic Attack (TIA) within 12 weeks of screening.
* History of syncope within the last 12 weeks prior to screening or sustained ventricular tachycardia without an implantable cardioverter-defibrillator.
* Moderate or severe aortic and/or mitral valve stenosis.
* Medically documented unstable angina, acute coronary syndrome (e.g., myocardial infarction, troponin-positive with symptoms of angina or unstable angina) within the last 8 weeks prior to start of screening.
* Medically documented ST-elevation myocardial infarction within 12 weeks of screening.
* Any tachycardia (inclusive of Atrial Fibrillation (AF) or atrial flutter) with a resting ventricular rate > 110 beats per minute at screening.
* For participants with a history of AF or atrial flutter, not on adequate anticoagulant therapy via non-vitamin K oral anticoagulants or warfarin if the CHA2DS2-VASc score is ≥ 2 in men or ≥ 3 in women or per local guidelines. Percutaneous occlusion of the left atrial appendage alone is not adequate.
* AF ablation within the last 12 weeks prior to screening or planned during the study duration.
* Symptomatic bradycardia or second (Mobitz Type II)- or third-degree heart block without a pacemaker.
* Cardiac surgery, coronary artery revascularization or indication for coronary artery revascularization, percutaneous coronary intervention, valve repair/replacement or valvuloplasty within 12 weeks prior to screening.
* Implantation of a Cardiac Resynchronization Therapy (CRT) device within 12 weeks prior to screening, or intent to implant a CRT device during the course of the study.
* Previous cardiac transplantation, or any use of mechanical circulatory support or similar device, or implantation expected after randomization.
* Receiving mechanical hemodynamic support or invasive mechanical ventilation within the last 8 weeks prior to screening.
* Receiving Intravenous (IV) inotropes or IV vasopressors within the last 8 weeks prior to screening.
* Receiving IV vasodilators within the last 4 weeks prior to screening.
* Receiving noninvasive mechanical ventilation within the last 4 weeks prior to screening. The use of noninvasive ventilation for sleep disordered breathing is permitted.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety - Cohort 1 | Study entry through week 52
  Incidence and severity of treatment emergent adverse events
Efficacy - Cohort 1 | Baseline through week 26
  Change in LVEF measured by 2D-TTE
Safety - Cohort 2 | Study entry through week 52
  Incidence and severity of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Locations (62):
- United States (51):
  - Site 121, Alexander City, Alabama
  - Site 130, Birmingham, Alabama
  - Site 139, Birmingham, Alabama
  - Site 138, Huntsville, Alabama
  - Site 111, Phoenix, Arizona
  - Site 127, Little Rock, Arkansas
  - Site 128, Huntington Beach, California
  - Site 157, Los Angeles, California
  - Site 158, Orange, California
  - Site 116, Pasadena, California
  - Site 129, Santa Maria, California
  - Site 102, Stanford, California
  - Site 113, Torrance, California
  - Site 133, Vista, California
  - Site 161, Coral Gables, Florida
  - Site 114, Hialeah, Florida
  - Site 162, Miami Lakes, Florida
  - Site 159, Naples, Florida
  - Site 136, Atlanta, Georgia
  - Site 143, Boise, Idaho
  - Site 160, Chicago, Illinois
  - Site 154, Park Ridge, Illinois
  - Site 137, Fort Wayne, Indiana
  - Site 112, Indianapolis, Indiana
  - Site 104, Covington, Louisiana
  - Site 118, Baltimore, Maryland
  - Site 119, Boston, Massachusetts
  - Site 122, Bloomfield Hills, Michigan
  - Site 150, Farmington Hills, Michigan
  - Site 107, Rochester, Minnesota
  - Site 106, St Louis, Missouri
  - Site 105, St Louis, Missouri
  - Site 144, Brick, New Jersey
  - Site 153, Valhalla, New York
  - Site 152, Asheville, North Carolina
  - Site 109, Cary, North Carolina
  - Site 140, Charlotte, North Carolina
  - Site 145, Durham, North Carolina
  - Site 117, Cincinnati, Ohio
  - Site 100, Cleveland, Ohio
  - Site 135, Oklahoma City, Oklahoma
  - Site 101, Portland, Oregon
  - Site 155, York, Pennsylvania
  - Site 110, Dallas, Texas
  - Site 115, Dallas, Texas
  - Site 103, Houston, Texas
  - Site 149, Tomball, Texas
  - Site 148, Arlington, Virginia
  - Site 123, Falls Church, Virginia
  - Site 126, Norfolk, Virginia
  - Site 163, Vienna, Virginia
- Canada (4):
  - Site 202, Winnepeg, Manitoba
  - Site 203, Brampton, Ontario
  - Site 200, Chicoutimi, Quebec
  - Site 201, Trois-Rivières, Quebec
- China (6):
  - Site 305, Changsha, Hunan
  - Site 303, Nanjing, Jiangsu
  - Site 306, Jining, Shandong
  - Site 301, Chengdu, Sichuan
  - Site 300, Beijing
  - Site 304, Chongqing
- Site 156, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No